CLINICAL TRIAL: NCT01128296
Title: Phase I/II Study of Preoperative Gemcitabine in Combination With Oral Hydroxychloroquine (GcHc) in Subjects With High Risk Stage IIb or III Adenocarcinoma of the Pancreas
Brief Title: Study of Pre-surgery Gemcitabine + Hydroxychloroquine (GcHc) in Stage IIb or III Adenocarcinoma of the Pancreas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amer Zureikat (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Amer Zureikat, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-122; PO1101944
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Cancer
Keywords: high risk stage IIb or III adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Hydroxychloroquine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydroxychloroquine + Gemcitabine (HcGc) (Experimental): Hydroxychloroquine orally twice daily in combination with gemcitabine for 31 days prior to surgical resection
  Interventions: Drug: Hydroxychloroquine; Drug: Gemcitabine

INTERVENTIONS:
Drug: Hydroxychloroquine — Oral dosing daily starting at 48 hours before first dose of gemcitabine (starting on Day -2) and for a total of 31 days (ending on Day 29), prior to surgical resection. Capsules are available in 200 mg strengths. Daily doses are 200, 400, 600, 800, 1000, or 1200 mg, and will be administered BID for doses above 200 mg.
  Other Names: Plaquenil
Drug: Gemcitabine — Intravenous administration on Days 1 and 15, with the infusion given at the fixed dose rate of 10mg/m2/min (e.g. 150 min for a 1500 mg/m2 dose).
  Other Names: Gemzar

SUMMARY:
The primary goal of the research study is to determine whether treating pancreatic cancer patients with hydroxychloroquine in combination with gemcitabine before surgery is safe. The secondary goal is to determine if this new treatment regimen can effectively treat pancreatic cancer. This study will test the safety and efficacy of this combination in two parts, or phases.

DETAILED DESCRIPTION:
This is a phase I/II trial designed to assess the safety, tolerability and efficacy of neoadjuvant oral hydroxychloroquine (Plaquenil®) in combination with FDR gemcitabine in subjects with high risk IIb or III adenocarcinoma of the pancreas. Eligible subjects will be administered hydroxychloroquine orally once or twice daily (depending on dose) in combination with FDR gemcitabine (on days 1 and 15) for 31 days prior to surgical resection. Dose escalations of hydroxychloroquine will proceed using Storer's Up-and-Down algorithm D. Subjects will be monitored for side effects and tolerability of the drug. Pre- and post-treatment PET scans will be the primary means to assess response to therapy. Resected tumors will also be assessed for evidence of inhibition of autophagy as well as histopathologic response and margin negative resection and number of positive lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with biopsy-proven adenocarcinoma of the pancreas
* staged by IIb or greater by by EUS, or tumor greater than 2.6 cm on EUS or pancreatic protocol helical CT scan demonstrating venous involvement
* Karnofsky performance status >/= 70.
* No active second malignancy except for basal cell carcinoma of the skin
* Normal renal, hepatic, and hematologic function at the time of enrollment as evidenced by:

  * Serum creatinine level ≤1.5 the upper limits of normal
  * Serum total bilirubin level ≤1.5 X ULN
* White blood cell count >/= 3.5x109/ml per ml and platelet count ≥ 100x109 per ml
* Age >18 years.
* For subjects with obstructive jaundice, the biliary tract must be drained with a temporary plastic or a short permanent metallic biliary stent.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects deemed surgically unresectable or subjects unwilling to undergo surgical resection.
* Subjects who have received chemotherapy within 12 months prior to study entry.
* Prior use of radiotherapy or investigational agents for pancreatic cancer.
* Any evidence of metastasis to distant organs (liver, lung, peritoneum).
* Symptomatic or endoscopic evidence of gastric outlet obstruction
* Concurrent malignancies with evidence of active or measurable disease except basal cell carcinoma of the skin
* Inability to adhere to study and/or follow-up procedures
* History of allergic reactions or hypersensitivity to the study drugs (hydroxychloroquine, gemcitabine).
* Other concurrent experimental therapy.
* The effects of HCQ, and gemcitabine on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. All females of childbearing potential must have a blood test or urine study within two weeks prior to registration to rule out pregnancy. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately. If a man impregnates a woman while participating in this study, he should inform his treating physician immediately as well.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with bone marrow-suppressive therapy, HIV-positive patients are excluded from the study. For patients receiving combination anti-retroviral therapy, the potential impact of pharmacokinetic interactions with HCQ and gemcitabine is unknown. Appropriate studies may be undertaken in patients with HIV and those receiving combination anti-retroviral therapy in the future.
* Due to the risk of disease exacerbation, patients with porphyria are ineligible.
* Patients with psoriasis are ineligible unless the disease is well controlled and they are under the care of a specialist who agrees to monitor the patient for exacerbations.
* Patients requiring the use of enzyme-inducing anti-epileptic medication that includes: phenytoin, carbamazepine, phenobarbital, primidone or oxcarbazepine are excluded.
* Patients with previously documented macular degeneration or diabetic retinopathy are excluded.
* Baseline EKG with QTc >470 msec (including subjects on medication). Subjects with ventricular pacemaker for whom QT interval is not measurable will be eligible on a case-by-case basis.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Zeh, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPCI/UPMC Cancer Centers, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Boone BA, Murthy P, Miller-Ocuin J, Doerfler WR, Ellis JT, Liang X, Ross MA, Wallace CT, Sperry JL, Lotze MT, Neal MD, Zeh HJ 3rd. Chloroquine reduces hypercoagulability in pancreatic cancer through inhibition of neutrophil extracellular traps. BMC Cancer. 2018 Jun 22;18(1):678. doi: 10.1186/s12885-018-4584-2. PMID 29929491

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 enrolled
  2 participants withdrew prior to treatment
  1 participants removed from protocol after the first dose of gemcitabine due to cerebrovascular accident unrelated to study drug
  1 patient removed from protocol due to allergic rash likely related to gemcitabine
  31 participants remained to receive gemcitabine + HCQ treatment
Groups:
- Preoperative Gemcitabine (1500 mg/m^2) + HCQ (200 mg/Day): Participants wtih pancreatic adenocarcinoma treated with two doses of fixed dose gemcitabine (1500 mg/m^2) administered (study days 3 and 17) in combination with oral HCQ dose of 200 mg/day taken for 31 consecutive days until the day of surgery.
- Preoperative Gemcitabine (1500 mg/m^2) + HCQ (400 mg/Day): Participants wtih pancreatic adenocarcinoma treated with two doses of fixed dose gemcitabine (1500 mg/m^2) administered (study days 3 and 17) in combination with oral HCQ dose of 400 mg/day taken for 31 consecutive days until the day of surgery.
- Preoperative Gemcitabine (1500 mg/m^2) + HCQ (600 mg/Day): Participants wtih pancreatic adenocarcinoma treated with two doses of fixed dose gemcitabine (1500 mg/m^2) administered (study days 3 and 17) in combination with oral HCQ dose of 600 mg/day taken for 31 consecutive days until the day of surgery.
- Preoperative Gemcitabine (1500 mg/m^2) + HCQ (800 mg/Day): Participants wtih pancreatic adenocarcinoma treated with two doses of fixed dose gemcitabine (1500 mg/m^2) administered (study days 3 and 17) in combination with oral HCQ dose of 800 mg/day taken for 31 consecutive days until the day of surgery.
- Preoperative Gemcitabine (1500 mg/m^2) + HCQ (1000 mg/Day): Participants wtih pancreatic adenocarcinoma treated with two doses of fixed dose gemcitabine (1500 mg/m^2) administered (study days 3 and 17) in combination with oral HCQ dose of 1000 mg/day taken for 31 consecutive days until the day of surgery.
- Preoperative Gemcitabine (1500 mg/m^2) + HCQ (1200 mg/Day): Participants wtih pancreatic adenocarcinoma treated with two doses of fixed dose gemcitabine (1500 mg/m^2) administered (study days 3 and 17) in combination with oral HCQ dose of 1200 mg/day taken for 31 consecutive days until the day of surgery.
Period: Overall Study
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (200 mg/Day) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (400 mg/Day) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (600 mg/Day) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (800 mg/Day) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (1000 mg/Day) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (1200 mg/Day)
Started | 1 | 1 | 1 | 1 | 1 | 26
Completed | 1 | 1 | 1 | 1 | 1 | 21
Not Completed | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day): Participants wtih pancreatic adenocarcinoma treated with two doses of fixed dose gemcitabine (1500 mg/m^2) administered (study days 3 and 17) in combination with oral HCQ (maximum dose of 1200 mg/day) taken for 31 consecutive days until the day of surgery.
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day)
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced a Dose Limiting Toxicity (DLT)
Description: Number of Participants at each dose level of HCQ that experienced a Dose Limiting Toxicity (DLT).
Time Frame: Up to 31 days
Population: Observed for dose-limiting toxicities or treatment delays attributed to HCQ to determine the maximum tolerated dose.
Measure: Number; unit: participants
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (200 mg/Day) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (400 mg/Day) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (600 mg/Day) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (800 mg/Day) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (1000 mg/Day) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (1200 mg/Day)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 26
participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Disease-free Survival (DFS)
Description: Median number of months of disease-free survival for participants receiving study treatment.
Time Frame: Up to 30 months
Population: Participants that completed more than 80 % of the intended dose of HCQ.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Preoperative Gemcitabine (1500 mg/m^2) + HCQ (1200 mg/Day): Participants with pancreatic adenocarcinoma treated with two doses of fixed dose gemcitabine (1500 mg/m^2) administered (study days 3 and 17) in combination with oral HCQ (1200 mg/day) taken for 31 consecutive days until the day of surgery.
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (1200 mg/Day)
Number analyzed (Participants) | 31
months | 11.97 [7.27 to 22.43]

3. Secondary Outcome: Overall Survival (OS)
Description: Median number of months of overall survival for participants receiving study treatment.
Time Frame: Up to 35 months
Population: Participants that completed more than 80% of the intended dose of HCQ.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day)
Number analyzed (Participants) | 31
months | 34.83 [11.57 to NA] — Upper bound of CI not reached due to too few events.

4. Secondary Outcome: Disease-free Survival (DFS) by Response to HCQ Treatment
Description: Median number of months of disease-free survival in participants who did and did not experience response to HCQ treatment. Patients who had >51 % increase in their LC3-II staining were classified as having a response to HCQ.
Time Frame: Up to 30 months
Population: Subset of participants that completed more than 80% of the intended dose of HCQ treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day)
Number analyzed (Participants) | 17
months
  Response to HQC treatment | 15.03 [6.8 to NA] — Upper bound not reached due to too few events.
  No response to HQC treatment | 6.9 [0.2 to NA] — Upper bound not reached due to too few events.

5. Secondary Outcome: Overall Survival (OS) by Response to HCQ Treatment
Description: Median number of months of overall survival in participants who did and did not experience response to HCQ treatment. Patients who had >51 % increase in their LC3-II staining were classified as having a response to HCQ.
Time Frame: Up to 35 months
Population: Subset of participants that completed more than 80 % of the intended dose of HCQ.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day)
Number analyzed (Participants) | 17
months
  Response to HQC treatment | 34.83 [11.7 to NA] — Upper bound of CI not reached due to too few events.
  No response to HQC treatment | 10.83 [0.02 to NA] — Upper bound of CI not reached due to too few events.

6. Secondary Outcome: R0 Resection Rate
Description: Number of participants that underwent a resection with microscopically margin-negative resection in which no gross or microscopic tumor remains in the primary tumor bed (24) / number of that completed treatment (31)
Time Frame: Up to 30 months
Population: Participants that completed more than 80 % of the intended dose of HCQ.
Measure: Number; unit: percentage of participants
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day)
Number analyzed (Participants) | 31
percentage of participants | 77

7. Secondary Outcome: Disease-free Survival (DFS) by CA 19-9 Response
Description: Median number of months of disease-free survival for participants who experienced Ca 19-9 (surrogate biomarker) response (either an increase or decrease in Ca 19-9), or no Ca 19-9 response. Per participant increases in Ca 19-9 ranged from >0 to 225%. Per participant decreases in Ca 19-9 ranged from >0 to 100%.
Time Frame: Up to 30 months
Population: Analysis population included a total of 26 participants who received study treatment, who experienced either an increase or decrease in Ca 19-9, or no Ca 19-9 surrogate biomarker response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day)
Number analyzed (Participants) | 26
months
  Ca 19-9 Response | 21.4 [9.1 to 24.2]
  No Ca 19-9 Response | 6.9 [2.3 to 9.7]

8. Secondary Outcome: Overall Survival (OS) by CA 19-9 Response
Description: Median number of months of overall survival for participants who experienced Ca 19-9 (surrogate biomarker) response (either an increase or decrease in Ca 19-9), or, no Ca 19-9 response. Per participant increases in Ca 19-9 ranged from >0 to 225%. Per participant decreases in Ca 19-9 ranged from >0 to 100%.
Time Frame: Up to 35 months
Population: Analysis population included participants who received study treatment, who experienced either an increase or decrease in Ca 19-9, or no Ca 19-9 surrogate biomarker response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day)
Number analyzed (Participants) | 26
months
  Ca 19-9 Response (increase or decrease) | 34.8 [11.7 to NA] — Upper bound of CI not reached due to too few events.
  No Ca 19-9 Response | 8.8 [5.6 to NA] — Upper bound of CI not reached due to too few events.

9. Secondary Outcome: Disease-free Survival by p53 Genetic Status
Time Frame: Up to 35 months
Population: Participants that completed more than 80 % of the intended dose of HCQ.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day)
Number analyzed (Participants) | 31
months
  p53 WT | 21.4 [5.5 to NA] — Upper bound of CI not reached due to too few events.
  p53 Mutant | 11.8 [6.9 to NA] — Upper bound of CI not reached due to too few events.

10. Secondary Outcome: Overall Survival (OS) by p53 Mutant Status
Time Frame: Up to 35 months
Population: Participants that completed more than 80 % of the intended dose of HCQ.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day)
Number analyzed (Participants) | 31
months
  p53 WT | NA [5.5 to NA] — Median and Upper bound of CI not reached due to too few events.
  p53 Mutant | 26.1 [8.8 to NA] — Upper bound of CI not reached due to too few events.

ADVERSE EVENTS:
Arm/Group | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day)
Serious Adverse Events (participants affected / at risk) | 4/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day) (N=35)
Infection with Grade 3-4 neutrophils (ANC <1.0x10^9/L), Abdomen NOS (Infections and infestations) | 1
Infection with Grade 3-4 neutrophils (ANC <1.0x10^9/L), Biliary tree (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Urinary tract NOS (Infections and infestations) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative Gemcitabine (1500 mg/m^2) + HCQ (≤1200 mg/Day) (N=35)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6
Platelets (Blood and lymphatic system disorders) | 10
Hemoglobin (Blood and lymphatic system disorders) | 23
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2
Weight loss (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 13
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 4
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 5
Distension/bloating, abdominal (Gastrointestinal disorders) | 2
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Anorexia (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 17
Hepatobiliary/Pancreas - Other (Specify, __) (Hepatobiliary disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2
Creatinine (Metabolism and nutrition disorders) | 2
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6
Alkaline phosphatase (Metabolism and nutrition disorders) | 9
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 11
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 12
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 14
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 17
Mood alteration, Anxiety (Nervous system disorders) | 2
Pain - Other (Specify, __) (General disorders) | 2
Pain, Abdomen NOS (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes